CLINICAL TRIAL: NCT02067962
Title: Identification of Genes Involved in Juvenile Idiopathic Arthritis by Wholel Exome Sequencing
Acronym: GenesinJIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9258
Record Dates: First submitted 2014-02-13; First posted 2014-02-20 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Arthritis, Juvenile Rheumatoid
Keywords: Juvenile idiopathic arhtritis; JIA; Gene identification; Whole exome sequencing; Next generation sequencing; Identification of molecular basis; Acceptation of both parents to participate to the study
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Juvenile idiopathic arthritis. (Other): Blood sample
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Blood sample

SUMMARY:
Juvenile idiopathic arthritis (JIA) is considered to be a multifactorial disease caused by a combination of environmental factors and predisposing genetic factors. Twins studies found a strong heritability (strong genetic factors) but genetic studies such association studies of large cohorts of patient (GWAS or Genome Wide Association Study) have elucidated less than 20 % of the genetic basis of JIA. The vision of the genetics of multifactorial diseases has recently changed revealing a large clinical and genetic heterogeneity of these diseases. Indeed, the advent of next-generation sequencing identified non-multifactorial genetic hereditary disease related to mutations in genes having strong effect on the onset of the disease without real impact of environmental factors among the so called "multifactorial diseases" (Parkinson's, diabetes, osteoarthritis, Alzheimer's, hypertension ...)The investigators propose to study 30 families with several forms of JIA by next-generation sequencing. Identifying the genetic basis of JIA in these families will help to better understand the physiopathology of this disease and may help to the identification of novel therapeutic targets for other patients with JIA.

ELIGIBILITY:
Inclusion Criteria:

* AJI oligoarticular form <4 joints
* AJI Polyarticular form> 4 joints
* AJI Forms systemic arthritis
* duration For more than six weeks
* Onset of symptoms before the age of 16 years
* Or rheumatoid factor or ANA + or CCP +Acceptation of both parenth to participate to the research and to perfom blood samples for genetic studies

Exclusion Criteria:

* The (the) patient (e) is under tutorship or curatorship
* The (the) patient (e) is under judicial protection
* The (the) patient (e), or his parents, refuses to sign the consent
* It is impossible to give (the) patient (e) information lit
* JIA spondyloarthropathies such
* JIA type psoriatic arthritis or enthesopathy
* JIA not classifiable

Ages: 1 Month to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03-05 (Actual); Primary Completion 2014-09-24 (Actual); Study Completion 2015-06-24 (Actual)

PRIMARY OUTCOMES:
Identification of new genes by Next Generation Squencing (NGS) | 1 day
  Identification of new genes by Next Generation Squencing (NGS) in order to propose a new classification for prognosis and therapeutic orientation

CONTACTS AND LOCATIONS:
Overall Officials: David DG GENEVIEVE, PU-PH, Principal Investigator — Montpellier University Hospital

REFERENCES:
- [Derived] Grandemange S, Sanchez E, Louis-Plence P, Tran Mau-Them F, Bessis D, Coubes C, Frouin E, Seyger M, Girard M, Puechberty J, Costes V, Rodiere M, Carbasse A, Jeziorski E, Portales P, Sarrabay G, Mondain M, Jorgensen C, Apparailly F, Hoppenreijs E, Touitou I, Genevieve D. A new autoinflammatory and autoimmune syndrome associated with NLRP1 mutations: NAIAD (NLRP1-associated autoinflammation with arthritis and dyskeratosis). Ann Rheum Dis. 2017 Jul;76(7):1191-1198. doi: 10.1136/annrheumdis-2016-210021. Epub 2016 Dec 13. PMID 27965258